CLINICAL TRIAL: NCT07361003
Title: A Phase Ib/III Study of Suvemcitug Plus Trifluridine/Tipiracil Tablets (FTD/TPI) Versus Placebo Plus Trifluridine/Tipiracil Tablets in Participants With Refractory Metastatic Colorectal Cancer
Brief Title: A Phase Ib/III Study of Suvemcitug Plus FTD/TPI in Participants With Refractory Metastatic Colorectal Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Jiangsu Simcere Pharmaceutical Co., Ltd. (Industry)
Collaborators: Jiangsu Simcere Biologics Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SIM0063-302; CTR20254831 (Registry Identifier: Center for drug Evaluation, NMPA)
Record Dates: First submitted 2025-09-30; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-12

CONDITIONS: Refractory Metastatic Colorectal Cancer
Keywords: refractory metastatic colorectal cancer; Suvemcitug; trifluridine/tipiracil
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Trifluridine; tipiracil

STUDY DESIGN:
Intervention Model Description: This study is divided into two parts: the first part (Phase Ib) is open-label, and the second part (Phase III) is a randomized double-blind study. This study is currently in the first part.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All study staff including the staff from sponsor, investigation site, contracted research organizations, blinded independent image review committee, site management organization and central lab are masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Suvemcitug+ trifluridine/tipiracil tablets (Experimental): Participants will receive Suvemcitug injection (at 1.5mg/kg for Phase Ib; and a recommended dose level based on Phase Ib result will be used for Phase III part) on Day 1 and Day 15 of each cycle (28 days), and trifluridine/tipiracil tablets at 35 mg/m² on day 1-5, 8-12 of each cycle (28 days), until disease progression, intolerable adverse event, participant withdrawal, or meet other discontinuation criteria as described by the protocol.
  Interventions: Drug: Suvemcitug injection, trifluridine/tipiracil tablets
- Placebo+ trifluridine/tipiracil tablets (Placebo Comparator): Participants will receive Suvemcitug placebo injection on Day 1 and Day 15 of each cycle (28 days), and trifluridine/tipiracil tablets at 35 mg/m² on day 1-5, 8-12 of each cycle (28 days), until disease progression, intolerable adverse event, participant withdrawal, or meet other discontinuation criteria as described by the protocol.
  Interventions: Drug: Suvemcitug placebo injection, trifluridine/tipiracil tablets

INTERVENTIONS:
Drug: Suvemcitug injection, trifluridine/tipiracil tablets — Suvemcitug injection at 1.5mg/kg, Trifluridine/tipiracil tablets at 35 mg/m²
  Arms: Suvemcitug+ trifluridine/tipiracil tablets
Drug: Suvemcitug placebo injection, trifluridine/tipiracil tablets — Suvemcitug placebo injection, Trifluridine/tipiracil tablets at 35 mg/m².
  Arms: Placebo+ trifluridine/tipiracil tablets

SUMMARY:
The primary goal of Phase Ib Study is to evaluate the safety of Suvemcitug in combination with trifluridine/tipiracil tablets in colorectal cancer participants.

The primary goal of Phase III Study is to evaluate the efficacy of Suvemcitug in combination with trifluridine/tipiracil tablets in colorectal cancer participants. Researchers will compare Suvemcitug + trifluridine/tipiracil tablets with placebo (a look-alike substance that contains no drug)+ trifluridine/tipiracil tablets to see if Suvemcitug + trifluridine/tipiracil tablets works better in treating refractory metastatic colorectal cancer.

DETAILED DESCRIPTION:
The study will enroll approximately 464 participants (30 for Phase Ib and 434 for Phase III stage) with refractory metastatic colorectal cancer who have previously received fluorouracil, oxaliplatin, and irinotecan-based chemotherapy, and who have either previously received or are unsuitable for anti-vascular endothelial growth factor (VEGF) therapy or anti-epidermal growth factor receptor (EGFR) therapy (RAS wild-type).

For Phase Ib Study, all 30 participants will be receiving the treatment with Suvemcitug in combination with trifluridine/tipiracil tablets. For Phase III Study, approximately 434 participants will be randomly assigned in a 1:1 ratio to two groups. One group will receive treatment with Suvemcitug + trifluridine/tipiracil tablets. The other group will receive the treatment with placebo + trifluridine/tipiracil tablets.

All participants will receive study treatment until they meet the criteria for treatment discontinuation. During study treatment period, investigators will evaluate the efficacy, safety and participants' quality of life. After treatment discontinuation, investigators will continue to follow up for subsequent treatment and survival information until the criteria for study discontinuation are met.

By the end of study, for participants who are still receiving study treatment, if their efficacy evaluation result is stable or response and they are tolerant to the treatment, then after obtaining approval from health regulatory authorities and ethics committees, they can continue study treatment by joining another extension study or in other ways as discussed by the sponsor.

ELIGIBILITY:
Inclusion Criteria:

* 1. Confirmed by histological and/or cytological examination as unresectable metastatic colon or rectal adenocarcinoma;
* 2. At least one measurable tumor lesion (RECIST v1.1);
* 3. Previously received fluorouracil, oxaliplatin, and irinotecan based chemotherapy; had previously undergone or was unsuitable for anti-VEGF therapy. (For participants with RAS wild-type, had previously undergone or was unsuitable for anti-EGFR therapy.);
* 4. Refractory metastatic colorectal cancer having progressed on or are intolerant to the last systemic treatment;
* 5. Good organ and bone marrow function (no administration of hematopoietic growth factors, blood transfusion, or platelets within 14 days before screening hematology test);
* 6. RAS mutation status confirmed by testing tumor tissue and /or blood sample.

Exclusion Criteria:

* 1. Having a second active primary malignancy within the past 5 years;
* 2. Symptomatic central nervous system (CNS) metastases or CNS metastases requiring local CNS-directed therapy (e.g., radiotherapy or surgery) or corticosteroid treatment within 2 weeks prior to the first administration of the study treatment;
* 3. Any active infection requiring systemic treatment within 2 weeks prior to the initiation of the study treatment;
* 4. Pleural effusion, pericardial effusion, or ascites that is uncontrolled or has required drainage or medical intervention within 4 weeks prior to the first administration of the study treatment;
* 5. Received systemic immuno suppressive therapy within 4 weeks prior to randomization (excluding prophylactic use or chronic low-dose steroids [≤20 mg/day prednisone equivalent dose]);
* 6. Currently taking or has recently taken (within 10 days prior to the first dose) aspirin (>325 mg/day);
* 7. Active or chronic hepatitis B (HBsAg or HBcAb positive and HBV DNA≥2000 IU/mL or ≥10000 copies/mL) or hepatitis C infection (HCV antibody positive and HCV RNA≥ULN);
* 8. Clinically significant cardiovascular disease within 6 months prior to the first administration of the study treatment;symptomatic coronary artery disease requiring medication; arrhythmia requiring medication (excluding asymptomatic atrial fibrillation with controlled ventricular rate); QTcF interval >470 ms at rest state; or uncontrolled hypertension or pulmonary hypertension;
* 9. Known hereditary or acquired bleeding and thrombotic tendencies (e.g., hemophilia, coagulation disorders, thrombocytopenia, hypersplenism, etc.); clinically significant bleeding events, arterial or deep venous thrombotic events, or superficial venous thrombosis and intermuscular venous thrombosis requiring intervention within 6 months prior to enrollment;
* 10. Participants with proteinuria (urine protein >2+ found during screening examinations; or urine protein 2+ with 24-hour urine protein quantification ≥1g/24h);
* 11. Participants with a history of intestinal obstruction (including incomplete intestinal obstruction) within 1 month prior to enrollment; participants with a history of abdominal fistula, gastrointestinal perforation, or abdominal abscess.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 464 (Estimated)
Dates: Start 2025-11-12 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Phase Ib: dose limiting toxicity (DLT) | At the end of Cycle 1 (each cycle is 28 days)
Phase Ib: Adverse Events | From signing informed consent form until 28 days after the last dose of study treatment, up to about 18 months
  The incidence (number of participants) and severity of adverse events (AE) and serious adverse events (SAE) assessed by CTCAE v5.0
Phase Ib: Tolerance | From signing informed consent until 28 days after the last dose of study treatment, for up to 18 months
  Number of participants who experienced adverse event related dose interruption, dose reduction and treatment discontinuation as assessed by investigators.
Phase III: overall survival (OS) | For about 18 months from the randomization of the last participant
  OS is the time interval from the date of randomization to death from any cause.

SECONDARY OUTCOMES:
Suvemcitug Serum concentration change over time of all participants | For about 6 cycles, each cycle is 28 days.
  Area under the serum concentration versus time curve (AUC)
Peak Suvemcitug serum concentration (Cmax) of all participants | For about 6 cycles, each cycle is 28 days
The time taken to reach peak Suvemcitug concentration after administration (Tmax) | For about 6 cycles, each cycle is 28 days
The time required for Suvemcitug concentration in the serum to decrease by half (t1/2) | For about 6 cycles, each cycle is 28 days
Serum anti-drug antibody (ADA) incidence of Suvemcitug | For about 6 cycles, each cycle is 28 days
  The number of participants with anti-drug antibody (ADA) tested positive from blood
Serum anti-drug antibody (ADA) duration of Suvemcitug | For about 6 cycles, each cycle is 28 days
  Duration of ADA measures how long the antibody persists in the blood
Serum anti-drug antibody (ADA) titer of Suvemcitug | For about 6 cycles, each cycle is 28 days
  ADA titer measures how much anti-drug antibody is present in the blood
Objective Response Rate (ORR) of all participants | From the date when the first dose of Suvemcitug is administered until radiological progression, initiation of new anti-cancer therapy, death or withdrawal from study, whichever came first, assessed up to 18 months.
  Proportion of participants who have a complete or partial response relative to baseline as assessed according to RECIST 1.1 criteria
Duration of response (DoR) of all participants | From the date when the first dose of Suvemcitug is administered until radiological progression, initiation of new anti-cancer therapy, death or withdrawal from study, whichever came first, assessed up to 18 months
  Measured from the date of partial or complete response to therapy until the cancer progresses based on RECIST v1.1 criteria.
Disease control rate (DCR) of all participants | From the date when the first dose of Suvemcitug is administered until radiological progression, initiation of new anti-cancer therapy, death or withdrawal from study, whichever came first, assessed up to 18 months.
  Proportion of participants who have a complete or partial response, or stable disease relative to baseline as assessed according to RECIST 1.1 criteria
Progression free survival (PFS) of all participants | From the date when the first dose of Suvemcitug is administered until radiological progression, initiation of new anti-cancer therapy, death or withdrawal from study, whichever came first, assessed up to 18 months.
Phase Ib: overall survival (OS) | For about 18 months from the randomization of the last participant
  OS is the time interval from the date of randomization to death from any cause
Phase III: Adverse Events | From signing informed consent form until 28 days after the last dose of study treatment, for about 18 months.
  The incidence (number of participants) and severity of adverse events (AE) and serious adverse events (SAE) assessed by CTCAE v5.0
Phase III: quality of life - EORTC QLQ-C30 | Questionnaires will be collected from participants at baseline, and all efficacy evaluation visits, for up to 18 months
  Quality of life evaluated by participant reported questionnaires: European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire - Core 30 .
Phase III: quality of life - Euro Qol (EQ)-5D | Questionnaires will be collected from participants at baseline, and all efficacy evaluation visits, for up to 18 months
  Evaluated by participant reported questionnaires: EuroQol- 5 Dimension Questionnaire.

CONTACTS AND LOCATIONS:
Locations (6):
- China (6):
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Harbin Medical University University Cancer Hospital, Harbin, Heilongjiang
  - The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - Cancer Hospital of Shandong First Medical University, Jinan, Shandong
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality
  - The Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Undecided